CLINICAL TRIAL: NCT02315859
Title: Validation of New Non-Invasive Parameters of Diastolic Suction in the Left Ventricle
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Gottfried und Julia Bangerter- Rhyner-Stiftung, Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 089/14
Record Dates: First submitted 2014-12-02; First posted 2014-12-12 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Diastolic Heart Failure
Keywords: suction work
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: All patients

SUMMARY:
It is known that, at the end of the cardiac ejection period, potential energy is stored in elastic fibers of the heart, which promotes the suction of blood from the atria during early filling. The investigators have developed a new ultrasound-based method to quantify this suction effect. Here, it is necessary to reduce the complex 3-dimensional cardiac mechanics in a 1-dimensional (piston-like) pump system. In the study, several steps of model reduction will be tested. Each reduction is intended to allow non-invasive measurements to become increasingly simple and feasible at reduced echo quality. The reference method is the invasive data obtained from a pressure-volume conductance catheter. To increase the supply of potential energy in the elastic fibers, a substance (dobutamine) is administered for transient strengthening of the force of contraction.

Hypothesis: There is a good agreement between the new, non-invasive parameters and the invasive reference method for the quantification of the suction effect of the left ventricle, and the good correlation persists even with increasing model simplification.

DETAILED DESCRIPTION:
Background

1. Clinical Background: Heart failure is a widespread cause of morbidity and mortality worldwide. Despite their similar clinical manifestation, systolic and diastolic heart failure are two distinct entities that differ with regard to pathophysiology, diagnosis, prognosis and treatment.

Diastolic dysfunction occurs early in the onset of heart failure. In the past, diastolic dysfunction has often been defined per exclusionem as heart failure in the absence of evidence of systolic dysfunction. This definition may be appropriate for clinical diagnosis if concentric or eccentric LV hypertrophy co-exists, but it is physiologically misleading, since diastolic dysfunction continues to persist or even worsens with the onset of systolic dysfunction. It should be considered that symptoms in heart failure are more closely related to diastolic than to systolic dysfunction. Furthermore, also prognosis of heart failure seems to be more closely related to the underlying degree of diastolic rather than systolic dysfunction. Despite its clinical importance, however, large trials on treatment outcome for diastolic heart failure (such as the CHARM-preserved and PEP-CHF trials) are scarce and disappointing. Among numerous others, three important reasons for this data scarcity are: overestimation of end-point events in the power analyses of the respective trials, lack of therapeutic agents that specifically target diastolic dysfunction, and lack of simple echocardiographic parameters capable of measuring diastolic function independently from loading conditions. The latter will be addressed in the study presented here. As will be detailed below, early-diastolic function is inextricably linked to the end-systolic conditions of the ventricle. An echocardiographic parameter describing an early-diastolic mechanical event is therefore very likely to vary with changes in end-systolic conditions. The present study will investigate new parameters of early-diastolic function by provoking contractility changes.

1.2 Physiological Background: There is no doubt that the human heart is a suction-pump capable of aspirating blood before expelling. There is a concept of early-diastolic suction: systolic myocardial shortening is believed to store potential energy in elastic fibers and myocyte filaments that are released in early-diastole to produce a suction effect, thus contributing to quick LV filling.

In 1930, Katz et al. first published a study describing a suction phenomenon in an in-vitro preparation of an isolated beating turtle ventricle. They showed that the early-diastolic volume increase of the ventricle coincides with a pressure fall, which is consistent with the concept of suction. He concluded that contraction and relaxation alters the elastic state of the ventricle between two limits (end-systolic and -diastolic), and proposed a suction effect produced by elastic recoil. This view represented a paradigm change, as filling was previously considered the result of atrial pressure. If suction is defined according to Katz, i.e. filling during pressure decay, then it is observed in all ejecting hearts, regardless of contractility, end-systolic volume or filling pressure. This type of suction corresponds to what early physiologists may have called the ventricular filling 'vis a fronte': a filling mechanism generated by the heart. It constitutes a suction effect relative to the filling reservoir. It can occur as a result of both, elastic recoil and relaxation.

In a physically more stringent concept, suction is defined as filling at negative LV transmural pressure. According to this definition, the ventricular wall performs work to pull blood into the cavity. There are two important conditions for such a suction event. First, the end-systolic volume must be lower than the volume of elastic ventricular equilibrium, otherwise no elastic energy would be stored. Second, early diastolic relaxation must be quick enough to allow restoring forces to prevail over the vanishing active forces. The process of suction lasts until the equilibrium volume is reached. Atrial pressure then stretches the ventricle to a volume where a force balance between filling pressure and ventricular passive stress impedes any further flow (diasthasis). Diasthasis volume is probably higher than the elastic equilibrium volume, which is a ventricular material property. Because LV filling itself very quickly abolishes any negative transmural pressures, and the equilibrium volume of the LV is probably small, suction according to this definition has been measured almost exclusively under particular circumstances, such as in nearly empty ventricles (e.g. artificially low afterload), during artificial absence of filling, or during inotropic stimulation.

1.3 Concept of Testing New Parameters: In the current study, several steps of model reduction will be tested. Each reduction is intended to allow non-invasive measurements to become increasingly simple and feasible at reduced echo quality. The comparison with the gold standard will then reveal the costs of model reductions in terms of precision and predictive power. Since direct pressure measurements are not feasible non-invasively, some simplifications of the pump model are mandatory. The most useful is to reduce the heart to a 1-dimensional, piston-like pump system moving only in apico-basal direction (longitudinal function). In such a model, not only contractions, but also flow directions are longitudinal. The 1-dimensional Euler equation can then be used to calculate instantaneous atrio-ventricular pressure gradients from Color Doppler M-Mode echocardiograms. Similarly, apico-basal displacement of the 'piston' can easily be measured by M-Mode echocardiograms of the mitral annulus (mitral annular plane systolic excursion, MAPSE). When combined, the suction effect of the ventricle relative to the left atrium can be assessed. A further simplification consists of replacing MAPSE by the widely used Doppler tissue imaging (DTI) -parameters of systolic (s') and early-diastolic (e') velocity. The reference method of this study will consist of invasively measured suction work, against which the new parameters will directly be compared.

Objective

The study is performed to prospectively test novel, non-invasive parameters of early diastolic function with respect to their ability to quantify the physiological phenomenon of LV suction.

Hypothesis: The following parameters correlate significantly with LV suction work, but in descending order of magnitude (r2): absolute suction work from pressure/MAPSE, relative suction work from IVPG/MAPSE, e'/L0, e'/s', (at rest and under Dobutamin).

Methods

Reference for LV suction work: conductance-catheter is introduced through the aortic valve and placed along the longitudinal axis of the LV. Continuous conductance are transformed into LV volume data and simultaneous pressure measurements are performed.

Echo parameters:

IVPG (intraventricular pressure gradients)is calculated from Color-Doppler M-Mode echocardiograms. This imaging modality produces a color-coded, longitudinal forward-flow velocity profile (y-axis) over time (x-axis). Such velocity maps can then be processed to retrieve instantaneous pressure gradients between any two points on the longitudinal axis.

MAPSE (mitral annular plane systolic excursion)is performed with M-Mode echocardiogram of the septal and lateral mitral annulus.

Tissue velocity: peak systolic velocity (s') and the peak early-diastolic negative velocity (e')of septal and lateral mitral anulus are measured by pulsed-wave Doppler tissue imaging (DTI).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients referred to elective percutaneous coronary angiography
* Stable cardio-pulmonary conditions
* Sinus rhythm
* Written informed consent to participate to the study

Exclusion Criteria

* Patients referred to emergency coronary intervention
* 2. Prior myocardial infarction, wall-motion-abnormalities, stenosis ≥50%
* Prior cardiac surgery
* More than mild left-sided valve disease
* Documented pulmonary disease leading to dyspnea NYHA II or more, including history of asthma bronchiale
* Any restrictive LV filling pattern without eccentric LV hypertrophy, such as in infiltrative myocardial diseases
* Pericardial diseases, including prior pericardiotomy and pericardial effusions.
* Pacemaker, implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy device (CRT)
* Known adverse reactions to Dobutamin or Esmolol
* Women who are pregnant or breast feeding (β-HCG > 10 IU/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with a large variety of clinical conditions leading to dyspnea (for example hypertensive or hypertrophic heart disease, dilated cardiomyopathy), and where no significant coronary artery disease or regional wall-motion abnormalities are identified.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Composite outcome measure: absolute suction work using MAPSE (Mitral annular plane systolic excursion) and IVPG (Intraventricular pressure gradients) | During the cardiac catheterization: at rest, under Dobutamin 20ug/kg, under Dobutamin 40ug/kg (expected average duration of 20 minutes); no follow-up.

SECONDARY OUTCOMES:
Composite outcome measure: absolute suction work using MAPSE and catheter-derived invasive pressure | During the cardiac catheterization: at rest, under Dobutamin 20ug/kg, under Dobutamin 40ug/kg (expected average duration of 20 minutes); no follow-up.
Composite outcome measure: absolute suction work using impedance catheter-derived volumes and IVPG | During the cardiac catheterization: at rest, under Dobutamin 20ug/kg, under Dobutamin 40ug/kg (expected average duration of 20 minutes); no follow-up.
Absolute suction work using tissue velocities (e'/s') | During the cardiac catheterization: at rest, under Dobutamin 20ug/kg, under Dobutamin 40ug/kg (expected average duration of 20 minutes); no follow-up.
Absolute suction work using tissue velocities (s'/L0, L0 = end-systolic ventricular length) | During the cardiac catheterization: at rest, under Dobutamin 20ug/kg, under Dobutamin 40ug/kg (expected average duration of 20 minutes); no follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, Prof, Study Chair; Stefano de Marchi, MD, Principal Investigator — Departement of Cardiology, Bern University Hospital
Locations (1):
- Departement of Cardiology, Bern University Hospital, Bern, Switzerland